CLINICAL TRIAL: NCT06564688
Title: To Explore the Functional Connectivity Pattern of Cortical Swallowing Network in the Oral Phase of Post-stroke Dysphagia Based on Dynamic Causal Modelling
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian University of Traditional Chinese Medicine (Other)
Collaborators: Xiangyang Central Hospital, Affiliated Hospital of Hubei University of Arts and Science (Other Government)
Responsible Party: Principal Investigator, Qingqing Zhang, lecturer, Fujian University of Traditional Chinese Medicine
Other Study IDs: 2023KY-015-02
Record Dates: First submitted 2024-08-12; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Dysphagia After Stroke; Cortical Swallowing Network; Functional Magnetic Resonance Imaging; Oral Phase; Dynamic Causal Modelling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dysphagia in the oral phase after stroke: The swallowing function was assessed by swallowing related scale and the Videofluoroscopic Swallowing Study, and then functional magnetic resonance imaging was performed.
  Interventions: Diagnostic Test: Swallowing function test
- Without dysphagia after stroke: First, the swallowing function related scale was evaluated, and then the functional magnetic resonance imaging (fMRI) scan was performed.
  Interventions: Diagnostic Test: Swallowing function test
- Healthy controls: First, the swallowing function related scale was evaluated, and then the functional magnetic resonance imaging (fMRI) scan was performed.
  Interventions: Diagnostic Test: Swallowing function test

INTERVENTIONS:
Diagnostic Test: Swallowing function test — The oral function score assesses the oral functional performance of chewing in all participants.
  The Functional oral feeding Scale (FOIS) was used to assess the ability of all participants to eat.
  The standardized swallowing assessment (SSA) was used to assess the global swallowing function of all participants.

SUMMARY:
Swallowing activity in the oral phase is regulated by the cortical swallowing network, and the functional connectivity pattern of the cortical swallowing network is related to swallowing activity. The structural damage of the cortical swallowing network and abnormal activation of brain areas related to swallowing in post-stroke dysphagia affect swallowing activity. The recovery of dysphagia after stroke is related to the compensation of swallowing network in the contralateral hemisphere and different connectivity patterns of diseased brain areas, and the integrity of cortical swallowing network connectivity affects the sequence of oral swallowing activities. However, it is not clear how the functional connectivity patterns and interactions of brain regions of the cortical swallowing network related to oral swallowing activity change in patients with oral dysphagia after stroke.

DETAILED DESCRIPTION:
Swallowing is a complex movement consisting of sequential and ordered activation of swallowing muscles interconnected cortical areas that facilitate the complex communication of sensory inputs and motor outputs to control oral movements such as jaw or chewing.During the swallowing task, the cortical swallowing network collaborates with each other to regulate swallowing activity. The damage of the swallowing cortex can affect the coordination of muscle groups in the swallowing process. Compared with healthy people, stroke patients show disordered swallowing movements, which greatly increases the risk of aspiration. Different lesions and connectivity patterns of stroke can affect the prognosis of dysphagia after stroke.In stroke patients with dysphagia, functional brain networks associated with motor control of swallowing were found to be disrupted in acute stroke patients with dysphagia.The recovery of dysphagia after stroke is related to the compensation of swallowing network in the contralateral hemisphere and different connectivity patterns of diseased brain areas, and the integrity of cortical swallowing network connectivity affects the sequence of oral swallowing activities. However, it is not clear how the functional connectivity patterns and interactions of brain regions of the cortical swallowing network related to oral swallowing activity change in patients with oral dysphagia after stroke.The purpose of this study is to explore the specific brain regions that are related to the dynamic changes of the functional connectivity pattern of the cortical swallowing network and the neuroimaging representations of the interbrain interaction in the oral phase of patients with dysphagia after stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria of patients with post-stroke oral dysphagia:

   * Patients with dysphagia after first stroke, meeting the diagnostic criteria of stroke, and confirmed by brain CT or brain MRI;
   * Oral dysphagia caused by stroke;
   * FOIS level ≤ 5; WST level ≥3;
   * Those who can understand and carry out the simple instructions of the treatment staff and are willing to accept the examination and treatment;
   * Clear consciousness and stable vital signs;
   * Patients in the recovery stage with stroke course and dysphagia duration between 0 and 6 months;
   * Right-handed;
   * Voluntary participants with informed consent.
2. Inclusion criteria of patients without dysphagia after stroke:

   * Patients with first-ever stroke, meeting the diagnostic criteria of stroke, and confirmed by brain CT or brain MRI;
   * No dysphagia, FOIS level =7; WST level =1;
   * Those who can understand and carry out the simple instructions of the treatment staff and are willing to accept the examination and treatment;
   * Clear consciousness and stable vital signs;
   * Patients in the recovery stage with stroke duration between 0 and 6 months;
   * Right-handed;
   * Voluntary participants with informed consent.
3. Inclusion criteria of healthy control group:

   * Normal cognitive function and swallowing function, FOIS level =7; WST level =1;
   * Gender and age matched with patients with dysphagia in the oral phase after stroke;
   * Right-handed;
   * Voluntary participants with informed consent.

Exclusion Criteria:

* Dysphagia not caused by stroke or non-oral dysphagia;
* History of cerebral trauma, stroke, brain tumor, cerebrovascular, intracranial infection, Parkinson's disease, epilepsy, or other neurological or psychiatric diseases;
* Symptoms of severe aphasia, neglect, visual field defect and other cortical lesions; Patients with severe cognitive impairment or depression;
* Taking or within 2 weeks of taking drugs that affect the nervous system or psychoses;
* Patients with metal implants and/or spatial claustrophobia who are not suitable for MRI scanning;
* Visual/hearing disorders affecting training and assessment;
* Persons who are participating in other research trials that may influence the results of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three categories of population were included in this study: post-stroke dysphagia in the oral phase, post-stroke dysphagia without dysphagia, and healthy controls. The subjects with post-stroke dysphagia were mainly those with oral dysphagia caused by the first stroke, who were able to complete the assessment and scanning, and had no contraindications to MRI scanning. The course of post-stroke dysphagia was between 0 and 6 months. The subjects without dysphagia after stroke were free of swallowing dysfunction after first stroke, could complete the assessment and scan, the course of stroke was between 0 and 6 months, and there were no contraindications to MRI scanning. The healthy controls were healthy people with normal cognition, swallowing function, and no contraindications to MRI scanning.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Standard Swallowing Assessment (SSA) | Before fMRI scan
  The scale has a minimum score of 18 and a maximum score of 46, with higher scores indicating poorer swallowing function
Oral Functional Scale | Baseline
  The Oral Functional Scale is a tool used to assess the oral functional status of an individual, with higher scores indicating better oral function

SECONDARY OUTCOMES:
Functional Oral Intake Scale (FOIS) | Baseline
  The Functional Oral Intake Scale (FOIS) is a reliable and valid tool for assessing functional oral food and fluid intake in patients with oropharyngeal dysphagia (OD). Fois has seven levels, with higher levels indicating better swallowing function.

OTHER OUTCOMES:
Videofluoroscopicdysphagia scale（VDS） | Baseline
  The VDS scale should be evaluated by videofluoroscopic swallowing study. The VDS has a total of 14 items, including 2 dimensions (oral phase and phase). Scores range from 0 to 100, with higher scores indicating greater severity of dysphagia.
Water Swallowing Test (WST) | Baseline
  Water Swallow Test (WST) is a method to evaluate the swallowing function of patients by observing their swallowing movements and performance during drinking water.

IPD SHARING:
Plan to Share IPD: No